CLINICAL TRIAL: NCT01733407
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy of L-Serine in Subjects With Hereditary Sensory Neuropathy Type 1
Brief Title: L-Serine Supplementation in Hereditary Sensory Neuropathy Type 1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Florian Eichler, Assistant Professor of Neurology, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FD-R-04127-01
Record Dates: First submitted 2012-09-19; First posted 2012-11-27 (Estimated); Results first posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-08

CONDITIONS: Hereditary Sensory and Autonomic Neuropathy Type I
Keywords: inherited neuropathies
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies | interventions — Serine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar pill (Placebo Comparator): Placebo arm
  Interventions: Drug: placebo
- L-serine (Active Comparator): amino acid supplementation with L-serine
  Interventions: Drug: L-serine

INTERVENTIONS:
Drug: L-serine — 400mg/kg/d L-serine or placebo divided TID for year 1, then crossover of placebo arm so that all patients on 400mg/kg/d L-serine divided TID for year 2.
  Other Names: amino acid supplementation with L-serine
  Arms: L-serine
Drug: placebo — 400mg/kg/d divided TID for year 1 only.
  Other Names: sugar pill
  Arms: Sugar pill

SUMMARY:
In hereditary sensory and autonomic neuropathy type 1 (HSAN1) the investigators recently discovered the accumulation of two neurotoxic sphingolipids. It appears that these lipids arise as the mutant enzyme has a reduced affinity for its normal preferred substrate L-serine. The investigators now plan to perform a two year study of L-serine supplementation to correct the biochemistry and neurological disease in humans with HSAN1. In the course the investigators will also establish correlations between an existing neurological rating scale of sensory neuropathy and intraepidermal nerve fiber density.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
The study objective is to evaluate the efficacy of L-serine in subjects with hereditary sensory neuropathy type 1 (HSAN1). Hereditary sensory and autonomic neuropathy type I (HSAN1) is a progressive and debilitating illness for which currently no treatment exists. The investigators recently identified two novel deoxysphingoid bases (DSB) that accumulate in plasma of HSAN1 patients and mutant transgenic HSAN1 mice. The disease is caused by missense mutations in the SPTLC1 gene encoding a subunit of the enzyme serine palmitoyltransferase (SPT). In normal circumstances the SPT enzyme catalyzes the reaction of palmitoyl-CoA with serine to form sphinganine. The two newly identified DSB, deoxysphinganine and deoxymethylsphinganine, arise from condensation of palmitoyl-CoA with alanine and glycine respectively, suggesting that HSAN1 mutations alter amino acid selectivity of SPT. In support of this hypothesis the investigators have shown that levels of DSB in humans and mice can be lowered by supplementation with the enzyme's normal substrate, serine.

In this randomized, double-blind, placebo-controlled cross over study the investigators will enroll 20 research participants with HSAN1 with 10 subjects assigned to L-serine (400mg/kg/d) and 10 assigned to placebo who are each treated for 12 months. The 10 subjects assigned to placebo will then be crossed over to active L-serine for the remaining 12 months. The progression of HSAN1 will be measured by the change in an established clinical rating scale and measures of intraepidermal nerve fiber density (IENFD) on skin biopsy. L-serine levels will be measured using 24-hour pharmacokinetic blood sample at 12-month intervals. The investigators will assess the percentage of failures (clinical decline of > 1 point on CMTNS or > 30% decrease in IENFD) at 6 month intervals. Regardless of CMTNS score, all subjects who are on placebo for the first year will be switched to active study drug in year two.

After the 2 year period subjects will be given the option of being re-consented for the open label extension. All consented subjects will then be treated with L-serine (400 mg/kg/d) for an additional year.

ELIGIBILITY:
Inclusion Criteria:

* HSAN1 patients with prominent sensory loss with foot ulcers or shooting pains and con-firmed mutations in SPTLC1.
* Males and females of 18 years or older
* All patients will be able to provide informed consent and comply with oral dietary supple-mentation and study activities. Compliance with supplementation will be monitored through measurement of DSB levels.
* Subjects must not have taken L-serine for at least 30 days prior to randomization (L-serine-naïve subjects are permitted in the study).
* Women must not become pregnant for the duration of the study and must be willing to use two contraceptive therapies and have a negative pregnancy test throughout the course of the study.

Exclusion Criteria:

* Any cause of neuropathy other than HSAN1 (such as diabetes or drug-induced neuropathy), medical history of kidney stones, or history of poliomyelitis or radiotherapy.
* Pregnant women, breastfeeding, or not using adequate contraception; for women included, an accepted method of contraception will be used throughout the study.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Patients on blood-thinners such as warfarin (Coumadin) or heparin will not be biopsied until they have held the medication for 5 days. Following the biopsy they will resume the maintenance dose of their medication.
* Serious illness (requiring systemic treatment and/or hospitalization) until subject either completes therapy or is clinically stable on therapy, in the opinion of the site investigator, for at least 10 days prior to study entry.
* The presence of unstable psychiatric disease, cognitive impairment, or dementia that would impair ability of the subject to provide informed consent, according to PI judgment, or a history of active substance abuse within the prior year.
* Subjects who are non-ambulatory.
* Subjects with uncontrolled diabetes.
* Patients who are unable or unwilling to give consent will not be enrolled in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-09; Primary Completion 2016-05 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Florian S Eichler, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - UMass Medical Center, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garofalo K, Penno A, Schmidt BP, Lee HJ, Frosch MP, von Eckardstein A, Brown RH, Hornemann T, Eichler FS. Oral L-serine supplementation reduces production of neurotoxic deoxysphingolipids in mice and humans with hereditary sensory autonomic neuropathy type 1. J Clin Invest. 2011 Dec;121(12):4735-45. doi: 10.1172/JCI57549. PMID 22045570
- [Derived] Fridman V, Suriyanarayanan S, Novak P, David W, Macklin EA, McKenna-Yasek D, Walsh K, Aziz-Bose R, Oaklander AL, Brown R, Hornemann T, Eichler F. Randomized trial of l-serine in patients with hereditary sensory and autonomic neuropathy type 1. Neurology. 2019 Jan 22;92(4):e359-e370. doi: 10.1212/WNL.0000000000006811. Epub 2019 Jan 9. PMID 30626650

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sugar Pill | L-serine
Started | 9 | 9
Completed | 7 | 9
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | L-serine | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (16.9) | 45.8 (11.0) | 47.8 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 5 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 9 | 17
  Canada | 1 | 0 | 1
Charcot-Marie-Tooth Neuropathy Score [Mean (Standard Deviation); unit: scores on a scale] — The Charcot Marie Tooth Neuropathy Score (CMTNS) is a 36-point composite scoring assessment that assesses disease severity in neuropathies. It is composed of 9 items that evaluate functions related to disease progression including assessing sensory symptoms, motor symptoms, pinprick sensibility, vibration, leg strength, arm strength, and nerve conduction tests. Each item is scored from 0 to 4 with the lower scores representing less severe symptoms and higher scores representing more severe symptoms.The individual item scores are then totaled to provide a global measure of disease severity
  scores on a scale | 24.6 (7.0) | 20.6 (10.0) | 22.6 (8.6)

OUTCOME MEASURES:

1. Primary Outcome: Charcot Marie Tooth Neuropathy Score
Description: The Charcot Marie Tooth Neuropathy Score (CMTNS) is a 0 to 36 point composite scoring assessment that is used to measure disease severity in Charcot Marie Tooth Neuropathy and other sensory and motor neuropathies. The CMTNS is composed of 9 items that evaluate functions related to disease progression. These 9 parameters include reviewing sensory symptoms, motor symptoms (arms and legs), pinprick sensibility, vibration, leg strength, arm strength, and nerve conduction tests. Each item is scored from 0 to 4, with the lower scores representing less severe symptoms and higher scores representing more severe symptoms.The 9 individual item scores are then totaled to provide a global measure of disease severity. For example the lowest possible total score is 0 which represents an asymptomatic individual and the highest score possible is a 36 which represents an individual with severe disease progression. There are sub scores that can be assessed but sub scores were not utilized in this study
Time Frame: 48 Weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sugar Pill | L-serine
Number analyzed (Participants) | 9 | 9
scores on a scale | 25.67 (6.69) | 20.22 (10.10)

2. Secondary Outcome: Intraepidermal Nerve Fiber Density (IENFD)
Description: Counts of nerve fibers per unit area in skin biopsies
Time Frame: 48 Weeks
Measure: Mean (Standard Deviation); unit: nerve fibers per micrometer^2
Arm/Group | Sugar Pill | L-serine
Number analyzed (Participants) | 9 | 9
nerve fibers per micrometer^2
  Upper Thigh | 34.67 (35.12) | 49.56 (43.44)
  Lower Calf | 0.89 (2.67) | 13.89 (24.10)

3. Secondary Outcome: Autonomic Function Testing (AFT) Composite Autonomic Severity Score (CASS)
Description: Autonomic Function Testing (AFT) tests the effectiveness of your autonomic nervous system which regulates important functions such as blood pressure, heart rate, and respiration. AFT results are quantified using the composite autonomic severity score scale (CASS) which is a scale from 0 to 10 that is the sum of three sub scores (cardiovagal, adrenergic, and sudomotor). Cardiovagal is scored from 0 to 3, sudomotor is scored from 0 to 3, and adrenergic is scored from 0 to 4. The tests include deep breathing, Valsalva maneuver, head-up tilt, and a sweat test. The three subscores are then summed. This total represents the CASS which classifies autonomic function as normal functioning (total score 0), mild (total score 1-3), moderate (total score 4-6), or severe (total score 7-10).
Time Frame: 48 Weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sugar Pill | L-serine
Number analyzed (Participants) | 9 | 9
scores on a scale | 3.56 (1.24) | 2.22 (1.64)

4. Secondary Outcome: Nerve Conduction Testing
Description: Evaluates the functioning of electrical conduction of the motor and sensory nerves of the human body.
Time Frame: 48 Weeks
Measure: Mean (Standard Error); unit: microvolts
Arm/Group | Sugar Pill | L-serine
Number analyzed (Participants) | 9 | 9
microvolts
  Sensrory Right Median Amplitude | 1.34 (4.03) | 5.51 (9.27)
  Sensory Right Antebrach Amplitude | 2.31 (3.94) | 5.89 (9.54)
  Sensory Right Superficial Radial Amplitude | 4.56 (10.17) | 10.84 (20.11)
  Sensory Right Sural Amplitude | 0.52 (1.57) | 1.07 (2.61)
  Sensory Right Superficial Peroneal Amplitude | 0.00 (0.00) | 0.00 (0.00)
  Motor Right Median (Wrist) Amplitude | 3.34 (4.52) | 4.21 (4.29)
  Motor Right Ulnar (Wrist) Amplitude | 2.49 (3.60) | 4.37 (4.80)
  Motor Right Peroneal EDB (Ankle) Amplitude | 0.54 (1.52) | 0.24 (0.66)
  Motor Right Peroneal Tib (Below) Amplitude | 0.29 (0.47) | 1.39 (2.15)

5. Secondary Outcome: 1-deoxy-sphinganine
Description: Plasma levels of the deoxysphingoid lipid 1-deoxy-sphinganine measured by liquid chromatography/mass spectrometry after hydrolyzing the N-acyl and O-linked headgroups
Time Frame: 48 Weeks
Measure: Mean (Standard Deviation); unit: micromole per liter
Arm/Group | Sugar Pill | L-serine
Number analyzed (Participants) | 9 | 9
micromole per liter | 0.338 (0.191) | 0.112 (0.042)

6. Secondary Outcome: 1-deoxy-sphingosine
Description: Plasma levels of the deoxysphingoid lipid 1-deoxy-sphingosine measured by liquid chromatography/mass spectrometry after hydrolyzing the N-acyl and O-linked headgroups
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: micromole per liter
Arm/Group | Sugar Pill | L-serine
Number analyzed (Participants) | 9 | 9
micromole per liter | 0.698 (0.306) | 0.337 (0.132)

ADVERSE EVENTS:
Arm/Group | Sugar Pill | L-serine
All-Cause Mortality (participants affected / at risk) | 1/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9 | 1/9
Other Adverse Events (participants affected / at risk) | 9/9 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill (N=9) | L-serine (N=9)
Esophageal Cancer (Gastrointestinal disorders) | 1 (1) | 0 (0) — Subject developed esophageal cancer
MRSA Staff Infection (Infections and infestations) | 0 (0) | 1 (1) — Hospitalized for MRSA Staff Infection
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill (N=9) | L-serine (N=9)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium Difficile Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Nail Infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal Infection (Infections and infestations) | 0 (0) | 1 (1)
Burns Second Degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Frostbite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood Sodium Decreased (Investigations) | 1 (1) | 0 (0)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Finger Amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Localized Infection (Infections and infestations) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes